CLINICAL TRIAL: NCT00390897
Title: Randomised Multicentre Phase IV Study to Compare Glivec® (Imatinib Mesylate, STI571) in Monotherapy Versus Glivec® in Combination With Interferon Alpha at Low Doses in the Treatment of Newly-Diagnosed Chronic-Phase Chronic Myeloid Leukaemia
Brief Title: Glivec® (Imatinib Mesylate, STI571) in Monotherapy Versus Glivec®-Interferon Alpha in the Treatment of Chronic-Phase Chronic Myeloid Leukaemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Pethema, pethema
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMC/PETHEMA; 03-0289
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Last update posted 2008-11-27 (Estimated); Status verified 2008-11

CONDITIONS: Chronic Myeloid Leukaemia
Keywords: chronic myeloid leukaemia; Glivec; Interferon
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; Interferons

INTERVENTIONS:
Drug: Glivec
Drug: Interferon

SUMMARY:
To compare the complete cytogenetic response rate in patients with newly-diagnosed chronic-phase chronic myeloid leukaemia treated with Glivec® alone or in combination with interferon at low doses

DETAILED DESCRIPTION:
Open, prospective, multicentre, phase IV, comparative and randomised study

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly-diagnosed chronic-phase Ph-positive chronic myeloid leukaemia (maximum 3 months as of the diagnosis of the disease, with the date of the cytogenetic study regarded as such).
2. Age between 18 and 72 years (both included).
3. Performance status < 2 on the ECOG scale (see Annex 3).
4. Secure written or oral informed consent in the presence of a witness and consent for biological samples (annexes 5 and 6).

Exclusion Criteria:

1. Criteria of acceleration or blastic crisis (see Annex 7).
2. When there is a compatible family donor in patients aged under 40 years or a non-relative donor in patients aged under 30 years (in whom allogenic transplant is still regarded as first-line treatment), the possibility of performing an allogenic transplant as first therapeutic option should be considered. In any case, as this aspect is still a matter of debate, it is left up to each group to take the relevant decision depending on the institution's policy.
3. Administration of other treatments before inclusion in the protocol (a maximum of 3 months of monotherapy with hydroxyurea is permitted).
4. Altered hepatic or renal function (SGOT, SGPT, total bilirubin and creatinine > 1.5 times the upper limit of normality).
5. Uncontrolled diseases, such as thyroidal dysfunction, diabetes mellitus, angina pectoralis, serious heart failure (functional class III/IV of the New York Heart Association classification), neuropsychiatric infection or disease (see annex 15).
6. Positive serology for HIV.
7. Record of cancer in the last 5 years (barring basal cell skin carcinoma and cervical carcinoma in situ).
8. Pregnancy or breastfeeding

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2003-07; Primary Completion 2006-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The fundamental objective of this study is to compare the therapeutic efficacy of Glivec® given in monotherapy (providing for dose scaling according to the response obtained at different periods of time from the beginning) in combination with standard in
The median survival of patients with CML is close to 7 years.
One year and a half after diagnosis, the rate of progression to the acceleration phase and blastic crisis is very low (3.3%) in patients treated with Glivec® as first line.
With the treatments available hitherto, the achievement of a major cytogenetic response and above all cytogenetic response translates into a prolongation of survival.
Therefore, taking into account that the rate of complete cytogenetic responses to Glivec® in newly-diagnosed CML is 76% after 18 months of treatment (see table I), the fundamental objective of the study will be to compare the rate of complete cytogenetic

SECONDARY OUTCOMES:
The time until complete cytogenetic responses are obtained
Rate of major cytogenetic responses
Rate of molecular responses
Time to the loss of cytogenetic, haematological or molecular response
Time to the progression of the disease to the phases of acceleration and blastic crisis (analysed according to intention to treat)
Survival (analysed according to intention to treat)
Haematological and non haematological tolerance and safety

CONTACTS AND LOCATIONS:
Overall Officials: Cervantes Francisco, Dr, Study Chair — Hospital Clinic of Barcelona
Locations (51):
- Spain (51):
  - Hospital Ntra. Sra. Sonsoles, Ávila, Avila
  - Hospital Son Dureta, Palma de Mallorca, Balearic Islands
  - Hospital Clínic, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Sant pau, Barcelona, Barcelona
  - Hospital Universitario "Germans Trias i Pujol", Barcelona, Barcelona
  - Hospital vall d'Hebrón, Barcelona, Barcelona
  - Institut Català d'oncología, Barcelona, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital Mútua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Complejo Hospitalario Reina Sofía, Córdoba, Córdoba
  - Hospital Ruiz de Alda, Granada, Granada
  - Hospital Juan Ramón Jiménez, Huelva, Huelva
  - Hospital Médico Quirúrgico Ciudad de Jaén, Jaén, Jaen
  - Hospital Juan Canalejo, A Coruña, La Coruña
  - Hospital Arnau de Vilanova, Lleida, Lleida
  - Hospital de Alcorcón, Alcorcón, Madrid
  - Clínica La Concepción, Madrid, Madrid
  - Clínica Puerta de Hierro, Madrid, Madrid
  - Hospital Clínico San Carlos de Madrid, Madrid, Madrid
  - Hospital de Fuenlabrada, Madrid, Madrid
  - Hospital Doce de Octubre, Madrid, Madrid
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario Princcipe de Asturias, Madrid, Madrid
  - Hospital Son Llatzer, Palma de Mallorca, Mallorca
  - Hospital Universitario Morales Meseguer, Murcia, Murcia, Murcia
  - . Hospital Clínico Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Carlos Haya, Málaga, Málaga
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital del Río Carrión, Palencia, Palencia
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clínico Universitario de Salamanca, Salamanca, Salamanca
  - Hospital General, Segovia, Segovia
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Joan XXIII, Tarragona, Tarragona
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - Hospital Clínico Universitario, Valencia, Valencia
  - Hospital dr. Peset, Valencia, Valencia
  - Hospital General Universitario, Valencia, Valencia
  - Hospital Universitario la Fe, Valencia, Valencia
  - Hospital Meixoeiro, Vigo, Vigo
  - Hospital Xeral, Vigo, Vigo
  - Hospital Virgen de la Concha, Zamora, Zamora
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital general de Jerez de la Frontera, Jerez de la Frontera
  - Hospital comarcal de Valdeorras, O'Barco de Valdeorras

REFERENCES:
- [Background] RUDKIN CT, HUNGERFORD DA, NOWELL PC. DNA CONTENTS OF CHROMOSOME PH1 AND CHROMOSOME 21 IN HUMAN CHRONIC GRANULOCYTIC LEUKEMIA. Science. 1964 Jun 5;144(3623):1229-31. doi: 10.1126/science.144.3623.1229. PMID 14150328
- [Background] Rowley JD. Letter: A new consistent chromosomal abnormality in chronic myelogenous leukaemia identified by quinacrine fluorescence and Giemsa staining. Nature. 1973 Jun 1;243(5405):290-3. doi: 10.1038/243290a0. No abstract available. PMID 4126434
- [Background] Heisterkamp N, Jenster G, ten Hoeve J, Zovich D, Pattengale PK, Groffen J. Acute leukaemia in bcr/abl transgenic mice. Nature. 1990 Mar 15;344(6263):251-3. doi: 10.1038/344251a0. PMID 2179728
- [Background] Daley GQ, Van Etten RA, Baltimore D. Induction of chronic myelogenous leukemia in mice by the P210bcr/abl gene of the Philadelphia chromosome. Science. 1990 Feb 16;247(4944):824-30. doi: 10.1126/science.2406902.
- [Background] Goldman JM, Szydlo R, Horowitz MM, Gale RP, Ash RC, Atkinson K, Dicke KA, Gluckman E, Herzig RH, Marmont A, et al. Choice of pretransplant treatment and timing of transplants for chronic myelogenous leukemia in chronic phase. Blood. 1993 Oct 1;82(7):2235-8. PMID 8400272
- [Background] Italian Cooperative Study Group on Chronic Myeloid Leukemia; Tura S, Baccarani M, Zuffa E, Russo D, Fanin R, Zaccaria A, Fiacchini M. Interferon alfa-2a as compared with conventional chemotherapy for the treatment of chronic myeloid leukemia. N Engl J Med. 1994 Mar 24;330(12):820-5. doi: 10.1056/NEJM199403243301204. PMID 8114834
- [Background] Druker BJ, Talpaz M, Resta DJ, Peng B, Buchdunger E, Ford JM, Lydon NB, Kantarjian H, Capdeville R, Ohno-Jones S, Sawyers CL. Efficacy and safety of a specific inhibitor of the BCR-ABL tyrosine kinase in chronic myeloid leukemia. N Engl J Med. 2001 Apr 5;344(14):1031-7. doi: 10.1056/NEJM200104053441401. PMID 11287972
- [Background] Savage DG, Antman KH. Imatinib mesylate--a new oral targeted therapy. N Engl J Med. 2002 Feb 28;346(9):683-93. doi: 10.1056/NEJMra013339. No abstract available. PMID 11870247
- [Background] Kantarjian H, Sawyers C, Hochhaus A, Guilhot F, Schiffer C, Gambacorti-Passerini C, Niederwieser D, Resta D, Capdeville R, Zoellner U, Talpaz M, Druker B, Goldman J, O'Brien SG, Russell N, Fischer T, Ottmann O, Cony-Makhoul P, Facon T, Stone R, Miller C, Tallman M, Brown R, Schuster M, Loughran T, Gratwohl A, Mandelli F, Saglio G, Lazzarino M, Russo D, Baccarani M, Morra E; International STI571 CML Study Group. Hematologic and cytogenetic responses to imatinib mesylate in chronic myelogenous leukemia. N Engl J Med. 2002 Feb 28;346(9):645-52. doi: 10.1056/NEJMoa011573. PMID 11870241
- [Background] O'Brien SG, Guilhot F, Larson RA, Gathmann I, Baccarani M, Cervantes F, Cornelissen JJ, Fischer T, Hochhaus A, Hughes T, Lechner K, Nielsen JL, Rousselot P, Reiffers J, Saglio G, Shepherd J, Simonsson B, Gratwohl A, Goldman JM, Kantarjian H, Taylor K, Verhoef G, Bolton AE, Capdeville R, Druker BJ; IRIS Investigators. Imatinib compared with interferon and low-dose cytarabine for newly diagnosed chronic-phase chronic myeloid leukemia. N Engl J Med. 2003 Mar 13;348(11):994-1004. doi: 10.1056/NEJMoa022457. PMID 12637609
- [Background] Kantarjian HM, Talpaz M, O'Brien S, Giles F, Garcia-Manero G, Faderl S, Thomas D, Shan J, Rios MB, Cortes J. Dose escalation of imatinib mesylate can overcome resistance to standard-dose therapy in patients with chronic myelogenous leukemia. Blood. 2003 Jan 15;101(2):473-5. doi: 10.1182/blood-2002-05-1451. Epub 2002 Sep 12. PMID 12393385
- [Background] Rea D, Legros L, Raffoux E, Thomas X, Turlure P, Maury S, Dupriez B, Pigneux A, Choufi B, Reman O, Stephane D, Royer B, Vigier M, Ojeda-Uribe M, Recher C, Dombret H, Huguet F, Rousselot P; Intergroupe Francais des Leucemies Myeloides Chronique; Group for Research in Adult Acute Lymphoblastic Leukemia. High-dose imatinib mesylate combined with vincristine and dexamethasone (DIV regimen) as induction therapy in patients with resistant Philadelphia-positive acute lymphoblastic leukemia and lymphoid blast crisis of chronic myeloid leukemia. Leukemia. 2006 Mar;20(3):400-3. doi: 10.1038/sj.leu.2404115. PMID 16437142
- [Background] Deng M, Daley GQ. Expression of interferon consensus sequence binding protein induces potent immunity against BCR/ABL-induced leukemia. Blood. 2001 Jun 1;97(11):3491-7. doi: 10.1182/blood.v97.11.3491. PMID 11369642
- [Background] Bhatia R, Wayner EA, McGlave PB, Verfaillie CM. Interferon-alpha restores normal adhesion of chronic myelogenous leukemia hematopoietic progenitors to bone marrow stroma by correcting impaired beta 1 integrin receptor function. J Clin Invest. 1994 Jul;94(1):384-91. doi: 10.1172/JCI117333. PMID 7518835
- [Background] Thiesing JT, Ohno-Jones S, Kolibaba KS, Druker BJ. Efficacy of STI571, an abl tyrosine kinase inhibitor, in conjunction with other antileukemic agents against bcr-abl-positive cells. Blood. 2000 Nov 1;96(9):3195-9. PMID 11050003
- [Background] Kano Y, Akutsu M, Tsunoda S, Mano H, Sato Y, Honma Y, Furukawa Y. In vitro cytotoxic effects of a tyrosine kinase inhibitor STI571 in combination with commonly used antileukemic agents. Blood. 2001 Apr 1;97(7):1999-2007. doi: 10.1182/blood.v97.7.1999. PMID 11264164
- [Background] Kontsioti F, Pappa V, Papasteriadis C, Economopulos T, Dervenoulas J, Papageorgiou E, Kalantzis D, Valsami S, Pappa M, Raptis S. In vitro effect of STI-571 in combination with A-interferon of the proliferation, differentiation and apoptosis of K562 cells. Hematol J 2002; suppl 1:980.
- [Background] O´Brien SG, Vallance SE, Craddock C, Holyoake TL, Goldman JM. PEGIntron and STI571 combination evaluation study (PISCES) in chronic phase chronic myeloid leukaemia. Blood 2001; suppl.:3512.
- [Background] Trabacchi E, Bassi S, Saglio G, Rege-cambrin G, Bonifazi F, De Vivo A, Testoni N, Martinelli G, Ruggeri D, Amabile M, Giannini B, Alberti D, Fincato GL, Tura S, Rosti G, Baccarani M. Pegylated recombinant interferon alfa 2b (PEGIntron) associated with imatinib mesylate (Glivec) in Ph chronic myeloid leukaemia (CML) in early chronic phase: a phase II study of the ICSG on CML. Hematol J 2002, suppl. :586
- [Background] O´Dwyer ME, Mauro MJ, Aust S, Kuyl J, PaquetteR, Sawyers C, Druker BJ. Ongoing evaluation of the combination of imatinib mesylate (Glivectm) with low dose interferon-alpha for the treatment of chronic phase CML. Hematol J 2002; suppl. : 990
- [Derived] Cervantes F, Lopez-Garrido P, Montero MI, Jonte F, Martinez J, Hernandez-Boluda JC, Calbacho M, Sureda A, Perez-Rus G, Nieto JB, Perez-Lopez C, Roman-Gomez J, Gonzalez M, Pereira A, Colomer D. Early intervention during imatinib therapy in patients with newly diagnosed chronic-phase chronic myeloid leukemia: a study of the Spanish PETHEMA group. Haematologica. 2010 Aug;95(8):1317-24. doi: 10.3324/haematol.2009.021154. Epub 2010 Mar 10. PMID 20220063
- See also: Spanish association of Haematology — http://www.aehh.org